CLINICAL TRIAL: NCT02724397
Title: Linked Color Imaging (LCI) and Magnifying Blue Laser Imaging (BLI) Versus Standard White Light for the Detection of Adenomas and Serrated Lesions in the Proximal Colon
Brief Title: Linked Color Imaging/Magnifying Blue Laser Imaging vs. White Light for Adenomas and Serrated Lesions in Proximal Colon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 307-LCI/BLI-002
Record Dates: First submitted 2016-03-18; First posted 2016-03-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Colon Cancer
Keywords: Colon cancer; Diagnosis; Adenoma; Serrated lesions
MeSH Terms: conditions — Colonic Neoplasms; Disease; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): (White endoscopy and then LCI/BLI) The patients will be evaluated by Standard White Light and then Linked Color Imaging/Magnifying Blue Laser Imaging (LCI/BLI).
  Interventions: Device: White endoscopy and then LCI/BLI
- Control group (Active Comparator): (LCI/BLI then white endoscopy) The patients will be evaluated by Linked Color Imaging/Magnifying Blue Laser Imaging (LCI/BLI) and then White Light Endoscopy.
  Interventions: Device: LCI/BLI then white endoscopy

INTERVENTIONS:
Device: LCI/BLI then white endoscopy — First use of Linked Color Imaging/Magnifying Blue Laser Imaging (LCI/BLI) and then White Light Endoscopy to detect colonic adenomas.
  Other Names: Linked Color Imaging/Magnifying Blue Laser Imaging (LCI/BLI)
  Arms: Control group
Device: White endoscopy and then LCI/BLI — First use of White Light Endoscopy and then Linked Color Imaging/Magnifying Blue Laser Imaging (LCI/BLI) to detect colonic adenomas.
  Other Names: Linked Color Imaging/Magnifying Blue Laser Imaging（LCI/BLI)
  Arms: Experimental group

SUMMARY:
Linked color imaging (LCI) and magnifying blue laser imaging (BLI) are two new imaging systems used in endoscopy which are recently developed. BLI was developed to compensate for the limitations of NBI. BLI shows a bright image of the digestive mucosa, enabling the detailed visualization of both the microstructure and microvasculature. However, BLI still is not able to obtain sufficient brightness for distant lesions. The newly developed LCI system (FUJIFILM Co.) creates clear and bright endoscopic images by using short-wavelength narrow-band laser light combined with white laser light on the basis of BLI technology. LCI makes red areas appear redder and white areas appear whiter. Thus, it is easier to recognize a slight difference in color of the mucosa. This is a study to determine if using LCI of the colon, rather than the usual white light on the colon, will improve the detection of flat adenomas and serrated polyps. The polyps are called serrated because of their appearance under the microscope after they have been removed. They tend to be located up high in the colon, far away from the rectum. They have been definitely shown to be a type of precancerous polyp and it is possible that using LCI will make it easier to see them, as they can be quite difficult to see with standard white light. LCI/BLI enables endoscopists to accurately describe the pit pattern of adenomas. By comparing White Light Endoscopy and LCI/BLI, it will show if there is any comparable advantage to using one or the other for lesion detection and assessment.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing the use of linked color imaging (LCI) and magnifying blue laser imaging (BLI) versus standard white light for the detection of serrated lesions in the proximal colon (the colon proximal to the splenic flexure). The proximal colon has large intestine and many folds which will lead missing flat lesions. Recent studies have indicated that colonoscopy is more effective in preventing cancer in the left side of the colon than the right side of the colon. The reasons for this difference may be partly biologic, in that a special group of polyps known as serrated polyps, particularly sessile serrated adenomas, are located primarily proximal to the splenic flexure. These lesions are endoscopically subtle in that they are often flat, have the same color as the surrounding mucosa, and are hard to differentiate from normal mucosa. LCI makes red areas appear redder and white areas appear whiter. Thus, it is easier to recognize a slight difference in color of the mucosa. This study will test whether LCI will increase the detection of serrated lesions in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

--Consecutive adult patients undergoing an outpatient colonoscopy

Exclusion Criteria:

* unable to provide informed consent
* had undergone prior resection of the colon
* inflammatory bowel disease
* familial adenomatous polyposis, Peutz-Jeghers syndrome or other polyposis syndromes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Proximal Serrated lesions and colorectal adenomas in proximal colon | 6 months
  Quantity of serrated lesions and colorectal adenomas found in the proximal colon during colonoscopy was recorded and compared.

SECONDARY OUTCOMES:
Improvement of histological diagnosis for serrated lesions and colorectal adenomas using LCI/BLI by comparing with that under white endoscopy | 3 months
  It is anticipated that the use of Linked Color Imaging (LCI) and Magnifying Blue Laser Imaging (BLI) will significantly improve the histological detection of colonic adenomas and serrated lesions when detected as opposed to White Light Endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, M.D., Ph.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sato R, Fujiya M, Watari J, Ueno N, Moriichi K, Kashima S, Maeda S, Ando K, Kawabata H, Sugiyama R, Nomura Y, Nata T, Itabashi K, Inaba Y, Okamoto K, Mizukami Y, Saitoh Y, Kohgo Y. The diagnostic accuracy of high-resolution endoscopy, autofluorescence imaging and narrow-band imaging for differentially diagnosing colon adenoma. Endoscopy. 2011 Oct;43(10):862-8. doi: 10.1055/s-0030-1256510. Epub 2011 Jul 5. PMID 21732270
- [Result] Rex DK, Clodfelter R, Rahmani F, Fatima H, James-Stevenson TN, Tang JC, Kim HN, McHenry L, Kahi CJ, Rogers NA, Helper DJ, Sagi SV, Kessler WR, Wo JM, Fischer M, Kwo PY. Narrow-band imaging versus white light for the detection of proximal colon serrated lesions: a randomized, controlled trial. Gastrointest Endosc. 2016 Jan;83(1):166-71. doi: 10.1016/j.gie.2015.03.1915. Epub 2015 May 5. PMID 25952085
- [Derived] Min M, Deng P, Zhang W, Sun X, Liu Y, Nong B. Comparison of linked color imaging and white-light colonoscopy for detection of colorectal polyps: a multicenter, randomized, crossover trial. Gastrointest Endosc. 2017 Oct;86(4):724-730. doi: 10.1016/j.gie.2017.02.035. Epub 2017 Mar 9. PMID 28286095